CLINICAL TRIAL: NCT07136285
Title: PIb/II, Open-label, Multicenter Study to Evaluate the Safety, Tolerability and Efficacy of I.V. Olvi-Vec Combined With Platinum Plus Etoposide in Patients With Advanced SCLC Who Are Platinum-recurrent or Platinum-refractory
Brief Title: Olvi-Vec Combined With Platinum Plus Etoposide Therapy in Patients With Late Phase SCLC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Newsoara HYK Biopharmaceutical (Shanghai) Co., Ltd. (Industry)
Collaborators: Genelux Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Olvi-Vec-SCLC-202
Record Dates: First submitted 2025-07-02; First posted 2025-08-22 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-06

CONDITIONS: SCLC, Extensive Stage
MeSH Terms: interventions — Platinum; Cisplatin; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental (Experimental): Olvi-Vec will be administered for 3 days in C1, then starting from C2, platinum (platinum (cisplatin or carboplatin)) and episode are administrated each 21 days till patients could not tolerate.
  Interventions: Drug: Olvi-Vec; Drug: platinum (cisplatin or carboplatin); Drug: Etoposide

INTERVENTIONS:
Drug: Olvi-Vec — Olvi-Vec will be administered to patient for 3 days during C1
Drug: platinum (cisplatin or carboplatin) — After completing the first cycle of treatment of Olvi-Vec (+21 days after the last dose), Platinum （Carboplatin or Cisplatin）will be administrated on D1,D2 and D3 each 21 days (dosage according to the label) from Cycle 2 until disease progression or intolerable toxicity occurred.
Drug: Etoposide — After completing the first cycle of treatment of Olvi-Vec (+21 days after the last dose), Etoposide will be administrated on D1,D2 and D3 each 21 days (dosage according to the label) from Cycle 2 until disease progression or intolerable toxicity occurred.

SUMMARY:
Oncolytic virus product named Olvi-Vec combined with Platinum plus Etoposide in patients with late phase SCLC

DETAILED DESCRIPTION:
Olvi-Vec is a genetic engineering modification of acne virus. GLP preclinical studies include the safety, pharmacology, and toxicology have been completed. Clinical studies exploring efficacy and safety in different types of tumor are ongoing.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and voluntarily sign an informed consent form.
* Age ≥ 18 years old, gender not limited.
* Small cell lung cancer confirmed by organization or cytology.
* After receiving platinum based chemotherapy regimens and/or immunotherapy, platinum based chemotherapy regimens and/or anlotinib, and other recommended treatments according to guidelines, disease progression or recurrence has occurred.
* There should be at least one measurable target lesion during the baseline period, according to RECIST 1.1 (if a lesion that has received radiation therapy has obvious evidence of disease progression after radiation therapy, it can be used as a target lesion).
* ECOG physical condition score 0 or 1.
* Have sufficient bone marrow, liver and kidney organ function-

Exclusion Criteria:

* Compound small cell lung cancer and transformed small cell lung cancer.
* Patients with brain metastases and neurological symptoms; Note: Subjects with previous imaging evidence of brain metastases who have undergone local treatment (such as radiotherapy or surgery) for intracranial metastases and have stable lesions for more than 28 days without symptoms can be enrolled.
* Other primary malignant tumors other than small cell lung cancer (excluding non melanoma skin cancer, breast cancer in situ, cervical cancer in situ, and superficial bladder cancer, or other cancers that have been effectively controlled in the past three years and have no evidence of disease recurrence) were previously or currently combined.
* Clinically significant cardiovascular diseases At the beginning of the study treatment, the toxicity associated with previous anti-tumor treatments did not recover to ≤ CTCAE grade 1, except for hair loss and peripheral neurotoxicity of CTCAE grade 2.
* Known HIV infection (HIV antibody positive), active hepatitis B and C patients.
* Receive chemotherapy, targeted therapy, radiotherapy, and biological therapy, with less than 4 weeks since the first administration in this study; Or have received local radiotherapy within 2 weeks.
* Having undergone major surgery or significant traumatic injury within 28 days prior to the first administration of the investigational drug -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate safety of Olvi-Vec in patients from day 1 to end of study | Interval between the date of enrollment and the date of withdraw and completion of study, up to a maximum of 2 years.
  Frequency and severity of adverse events measured according to NCI Common Toxicity Criteria Adverse Event (CTCAE), version 5.0

SECONDARY OUTCOMES:
Explore the dose limiting toxicity (DLTs) during day 1 to day 25 of treatment cycle 1 | Day 1 to day 25 of treatment cycle 1
  Olvi-Vec related Grade 3 or higher adverse events (AEs) which meets DLT criteria.
Objective Response Rate (ORR) | Interval between the date of enrollment and the date of withdraw and completion of study, up to a maximum of 2 years.
  ORR is proportion of subjects with complete response(CR) or partial response(PR). Tumor responses will be evaluated according to RECIST 1.1 criteria. Patients with no tumor assessment after baseline will be classified as non-responders.
Disease control rate (DCR) | Interval between the date of enrollment and the date of withdraw and completion of study, up to a maximum of 2 years.
  DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks) based on RECIST V1.1
Progression free survival (PFS) | Interval between the date of enrollment and the date of withdraw and completion of study, up to a maximum of 2 years.
  PFS is defined as the time from the date of first dosing till the first documentation of disease progression (per RECIST v1.1) assessed by the investigator or death due to any cause (whichever occurs first)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Shanghai chest hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No